CLINICAL TRIAL: NCT05615844
Title: A Randomized Controlled Trial Comparing Antibiotic Cement Bead Pouch Versus Negative Pressure Wound Therapy for the Management of Severe Open Tibia Fracture Wounds
Brief Title: Antibiotic Cement Bead Pouch Versus Negative Pressure Wound Therapy
Acronym: BeadsvsVac
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: McMaster University (Other); University of California, Irvine (Other)
Responsible Party: Principal Investigator, Mark Gage, Associate Professor, Department of Orthopaedics, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSU00222774
Record Dates: First submitted 2022-10-14; First posted 2022-11-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Open tíbia Fracture
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotic Cement Bead Pouch (Experimental): The antibiotic cement bead pouch involves placing temporary non-absorbable antibiotic-laden cement beads into the open fracture wound and sealing the wound with a large occlusive dressing for prophylaxis against bacteria.
  The antibiotic beads used will be prepared intraoperatively by the surgical team. The bead recipe will be comprised of a ratio of 2 grams of vancomycin, 2.4 grams of tobramycin, and 40g (one bag) of PMMA cement. The beads will be handmade and approximately 10-mm in diameter. The number of beads placed in the wound will be at the discretion of the treating surgeon based on recipient wound size. As commonly practiced, the antibiotic beads may be exchanged for new beads at each subsequent irrigation and debridement surgery. The number of beads, the number of replaced beads, and the removal of the antibiotic beads will be recorded.
  Interventions: Drug: Antibiotic Cement Bead Pouch
- Negative Pressure Wound Therapy (NPWT) (Active Comparator): The NPWT system is a sealed dressing placed over the open fracture wound that includes an occlusive plastic wound dressing connected to a vacuum pump, tubing, and a canister to collect fluid. The pump creates a vacuum seal and exerts negative pressure on the wound to remove fluid and maintain a sealed environment. NPWT promotes wound healing through four primary mechanisms: 1) wound shrinkage or macrodeformation; 2) microdeformation at the foam-wound surface interface; 3) fluid removal; and 4) stabilization of the wound environment.
  125 mmHg continuous negative pressure is the recommended NPWT device setting; however, the treating surgeon will be allowed to adjust these settings as clinically necessary.
  The frequency and timing of NPWT changes will also be at the surgeon's discretion but is expected to primarily coincide with the timing of repeat debridement, typically every 24-72 hours until definitive management has occurred.
  Interventions: Device: Negative Pressure Wound Therapy

INTERVENTIONS:
Drug: Antibiotic Cement Bead Pouch — The antibiotic bead pouch provides an antibiotic delivery mechanism. It is made by combining polymethyl methacrylate (PMMA) cement with generic forms of vancomycin and tobramycin powder.
  Arms: Antibiotic Cement Bead Pouch
Device: Negative Pressure Wound Therapy — Standard application of negative pressure wound therapy
  Arms: Negative Pressure Wound Therapy (NPWT)

SUMMARY:
The Beads vs Vac trial is a multi-centre randomized controlled trial of 312 participants with a severe open tibia fracture requiring multiple irrigation and debridement surgeries. Eligible participants will be randomized to receive either an antibiotic bead pouch or negative pressure wound therapy (NPWT) for their temporary open fracture wound management. Outcomes will be assessed at 6 weeks, 3 months, and 6 months post-surgery. The primary outcome will be a composite outcome to evaluate clinical status six months after randomization. Components of the composite outcome will be hierarchically assessed in the following order: 1) all-cause mortality, 2) injury-related amputation of the lower extremity, 3) unplanned reoperation to manage wound complications, infection, or delayed fracture healing, and 4) clinical fracture healing as assessed using the Functional IndeX for Trauma (FIX-IT) instrument. The secondary outcomes will independently assess the four components of the primary outcome. This is a Phase III trial.

DETAILED DESCRIPTION:
The primary objective of early open fracture management is to minimize the risk of complications. In severe cases, multiple irrigation and debridement surgeries are required to overcome the severe wound contamination, to reassess the evolving tissue injury, and/or to temporize and plan appropriate soft tissue coverage with a skin graft or muscle flap. When multiple irrigation and debridement surgeries are needed, there is uncertainty on how the open fracture wound should be managed between procedures. Negative pressure wound therapy (NPWT), commonly known as a Wound VAC, is the preferred method of open fracture wound management for most surgeons. Opponents of NPWT believe that NPWT desiccates the open fracture wound and rapidly removes any local antibiotics placed in the wound during surgery. Instead of using NPWT, they place temporary non-absorbable antibiotic-laden cement beads into the open fracture wound and seal it with a large occlusive dressing. This wound management strategy is known as an antibiotic cement bead pouch, or more commonly a Bead Pouch. Mounting evidence questions the effectiveness of NPWT to prevent open fracture complications. Additionally, emerging comparative studies suggest the antibiotic bead pouch may significantly reduce the risk of infection compared to NPWT. This trial seeks to fill this critical knowledge gap.

The primary objective of this trial is to determine if the antibiotic bead pouch, compared to NPWT application, is more effective at reducing open tibia fracture complications. The primary outcome will be a composite outcome to evaluate clinical status six months after randomization. Components of the composite outcome will be hierarchically assessed in the following order: 1) all-cause mortality, 2) injury-related amputation of the lower extremity, 3) unplanned reoperation to manage wound complications, infection, or delayed fracture healing, and 4) clinical fracture healing as assessed using the Functional IndeX for Trauma (FIX-IT) instrument. The secondary objectives will independently assess the four components of the primary outcome.

The trial population includes patients 18 years and older with a severe open tibia fracture requiring more than one irrigation and debridement and being treated with internal or external fixation for definitive fracture management. Patients who have contraindications to the NPWT or local intrawound antibiotics will be excluded.

312 participants will be randomized in a 1:1 ratio to receive either an intraoperative antibiotic bead pouch or negative pressure wound therapy (NPWT). Participants will receive their allocated wound management strategy at the conclusion of their first irrigation and debridement procedure. Participants will have follow-up assessments at 6 weeks, 3 months and 6 months post-fracture.

The primary outcome will be a composite outcome to evaluate clinical status six months after randomization. Components of the composite outcome will be hierarchically assessed in the following order: 1) all-cause mortality, 2) injury-related amputation of the lower extremity, 3) unplanned reoperation to manage wound complications, infection, or delayed fracture healing, and 4) clinical fracture healing as assessed using the Functional IndeX for Trauma (FIX-IT) instrument. The secondary outcomes will independently assess the four components of the primary outcome. An Adjudication Committee will review all primary and secondary endpoints and a Data Safety Monitoring Committee (DSMC) will review all safety events.

ELIGIBILITY:
The inclusion criteria are:

1. Patients 18 years of age or older.
2. Severe open tibia fracture requiring more than one irrigation and debridement procedure to treat the open fracture.
3. Planned internal or external fixation for definitive fracture management.
4. Formal surgical debridement within 72 hours of their injury.
5. Will have all planned fracture care surgeries performed by a participating surgeon or delegate.
6. Informed consent obtained.

The exclusion criteria are:

1. Due to the severity of injury, the treating surgeon does not believe limb salvage >6 months is likely to be successful based on the emergency department or initial intraoperative assessment (prior to enrolment and randomization).
2. Medical contraindication to antibiotic beads, including previously known allergies or sensitivities to vancomycin and/or tobramycin.
3. Medical or injury contraindication to NPWT. Injury contraindications could include situations in which the NPWT could not be placed over a vascular graft or exposed neurovascular structure.
4. Received previous surgical debridement or management of their fracture at a non-participating hospital or clinic (as applicable).
5. Chronic or acute infection at or near the fracture site at the time of initial fracture surgery.
6. Incarceration.
7. Women of child-bearing potential who are pregnant or intending to become pregnant within the next 6 months.
8. Currently enrolled in a study that does not permit co-enrollment.
9. Unable to obtain informed consent due to language barriers.
10. Anticipated problems, in the judgment of research personnel, with maintaining follow-up with the patient.
11. Prior enrollment in the trial.
12. Other reason to exclude the patient, as approved by the Methods Center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2023-11-05 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical status | 6 months
  Clinical status is a hierarchal composite of the following outcomes:
  i) all-cause mortality ii) amputation at the fracture location iii) unplanned reoperation to manage wound complications, an infection, or promote fracture healing, iv) clinical fracture healing assessed using the Functional IndeX for Trauma (FIX-IT) instrument.

SECONDARY OUTCOMES:
Mortality | 6 months
  All-cause mortality
Amputation | 6 months
  Injury-related amputation of the lower extremity
Unplanned reoperation(s) | 6 months
  Unplanned reoperation to manage wound complications, an infection, or promote fracture healing.
Clinical fracture healing | 6 months
  Clinical fracture healing assessed using the Functional IndeX for Trauma (FIX-IT) instrument.

CONTACTS AND LOCATIONS:
Locations (32):
- United States (27):
  - Dignity Health Chandler Regional Medical Center, Chandler, Arizona
  - University of California, Davis, Davis, California
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Maryland, R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - University of Maryland Capital Region Health, Largo, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Mississippi, University, Mississippi
  - Bryan Medical Center, Lincoln, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Sanford Medical Center, Fargo, North Dakota
  - University of Cincinnati, Cincinnati, Ohio
  - Bon Secours Mercy Health, Cincinnati, Ohio
  - Slocum Center, Eugene, Oregon
  - Ortegon Health & Science University, Portland, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Prisma Health - Midlands, Columbia, South Carolina
  - Prisma Health, Greenville, South Carolina
  - Sanford Health, Sioux Falls, South Dakota
  - University of Utah, Salt Lake City, Utah
  - Inova Fairfax, Falls Church, Virginia
  - University of Wisconsin, Madison, Wisconsin
- Canada (5):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - University of British Columbia, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario